CLINICAL TRIAL: NCT03540394
Title: Long Term Outcomes of Pediatric Compartment Syndrome
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Abdelrahman Lawendy, Orthopaedic Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 111865
Record Dates: First submitted 2018-05-03; First posted 2018-05-30 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Compartment Syndromes
MeSH Terms: conditions — Compartment Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to review the etiology, diagnostic criteria, complications and outcome of acute pediatric compartment syndrome identified at The Children's Hospital of Western Ontario (CHWO) . Follow up with patients treated for compartment syndrome by fasciotomy will assist in determining the long term effects of compartment syndrome and surgical procedures on the patient quality of life and return to level of function of the affected limb.

DETAILED DESCRIPTION:
Acute compartment syndrome (ACS) is caused by elevated pressure within a closed osseofascial compartment, leading to microvascular compromise and cell death. Without urgent decompression of the compartment, significant functional impairment and loss of limb may result. Compartment syndrome can be difficult to diagnose as there are a wide variety of causes, clinical manifestations, and no reliable objective test. The diagnosis in a pediatric population is further complicated when the patient has a decreased ability to communicate verbally, and/or is non-compliant with physical examination. CS pathophysiology indicates that such an increase in compartmental pressure leads to the loss of microvascular perfusion (ischemia), restricting oxygen and nutrient delivery to vital tissues, ultimately causing the permanent functional and physical loss of the limb. The basic principle of fasciotomy is the full and adequate decompression of the compartment of interest and is performed secondary to compartment syndrome. This can be achieved via a single or double incision approach with both methods appearing to be equally effective in reducing intercompartment pressure (ICP). Subsequent skin closure and/or coverage is performed only when all muscle groups are deemed viable. However, there are a number of coverage techniques described without a clear systematic approach based on objective outcomes. Currently, the only available treatment consists of restoration of blood flow by releasing the pressure by slicing open the skin and connective tissue overlying the muscle in a procedure called fasciotomy. This crude method may result in long-term muscle weakness and disfigurement, and does not treat the ischemic damage already caused by the trauma. Pressure release can be achieved via a single or double incision approach with both methods appearing to be equally effective in reducing ICP. Subsequent skin closure and/or coverage is performed only when all muscle groups are deemed viable. However, there are a number of coverage techniques described without a clear systematic approach based on objective outcomes.

ELIGIBILITY:
Inclusion Criteria:

* skeletally immature patients (i.e under 18 years of age) admitted to Childrens Hospital of Western Ontario (CHWO) between January 2007 and 2017
* diagnosed compartment syndrome development
* required surgical intervention in the form of a fasciotomy for compartment syndrome of either the upper or lower extremity

Exclusion Criteria:

* 18 years of age or greater
* no development of diagnosed compartment syndrome

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients admitted to CHWO between 2007 and 2017 who underwent a fasciotomy for compartment syndrome of either an upper or lower extremity
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Function (LEF) | 1 year
  Function of lower Limb
Upper Extremity functional Index (UEFI) | 1 year
  Function of upper limb

SECONDARY OUTCOMES:
EQ5D | 1 year
  Overall generic health status

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Mubarak SJ, Owen CA. Double-incision fasciotomy of the leg for decompression in compartment syndromes. J Bone Joint Surg Am. 1977 Mar;59(2):184-7. PMID 15455478
- [Background] Vitale GC, Richardson JD, George SM Jr, Miller FB. Fasciotomy for severe, blunt and penetrating trauma of the extremity. Surg Gynecol Obstet. 1988 May;166(5):397-401. PMID 3363458